CLINICAL TRIAL: NCT01391715
Title: Double-dose Rabeprazole Accelerates and Sustains the Control of Symptoms in Patients With NERD: a Randomized Controlled Trial
Brief Title: Double-dose Rabeprazole Accelerates and Sustains the Control of Symptoms in Patients With NERD
Acronym: DRNERD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: patients could not be recuited within study duration
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Eun Hee Seo, Fellow, Inje University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01July2011
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal reflux disease; Proton pump inhibitor; standard dose; Double dose
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double dose rabeprazole (Active Comparator): Rabeprazole 20m bid per day will be given for 2 weeks
  Interventions: Drug: rabeprazole
- standard dose rabeprazole (Placebo Comparator): rabeprazole 20mg per day will bi given for 2 weeks
  Interventions: Drug: standard dose rabeprazole

INTERVENTIONS:
Drug: rabeprazole — rabeprazole 20mg bid per day for 2 weeks
  Arms: Double dose rabeprazole
Drug: standard dose rabeprazole — rabeprazole 20mg qd per day for 2 weeks
  Arms: standard dose rabeprazole

SUMMARY:
To the best of our knowledge, there has been no randomized controlled trial to compare double dose PPI therapy with standard one dose PPI therapy for NERD patients. Thus, we hypothesize that a double dose PPI would accelerate and sustain the control of symptom in NERD patients.

DETAILED DESCRIPTION:
In Asian, the majority of GERD cases are cases of nonerosive reflux esophagitis(NERD). NERD is a difficult -to-treat acid reflux condition even with PPI compared to reflux esophagitis(RE). In addition, the quality of life of NERD patients is quite low, NERD patients need quicker and more effective treatment options. At present, PPI-based step-down treatment is recommended for GERD patients. Doubling th PPI dose has become a commonly practiced therapeutic strategy in patients with GERD who failed PPI once daily. In patients with symptomatic GERD who failed the one dose PPI can increase the rate of overall symptom improvement by 22-26%. There are various mechanisms for standard dose PPI failure in GERD patients. Esophageal hypersensitivity is likely the underlying mechanism in a significant number of patients. Patients with the sensitive esophagus (normal endoscopy and pH test but positive symptom index) were more likely to respond to PPI twice a day. It is thus of clinical interest to determine whether an increased dosage of PPI can achieve rapidly the control of symptoms for patient with NERD patients.

ELIGIBILITY:
Inclusion Criteria:

* heartburn and/or reflux at least twice weekly in the absence of visible esophageal mucosal breaks at endoscopy

Exclusion Criteria:

* pregnancy
* lactation
* Hx of gastric surgery
* Hx of gastric cancer or peptic ulcer
* major medical problems (including CHF, renal failure, COPD, asthma, liver cirrhosis)
* severe systemic illness
* Hx of malignancy, allergy Hx to rabeprazole
* patients who had taken antibiotics
* antisecretory agents including H2-blocker
* PPI within 4 weeks before endoscopy
* current usage of steroids, NSAIDs, aspirin, anticoagulant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
symptom improvement at 2 week after double dose rabeprazole treatment | Two weeks
  symptom improvement according to FSSG(the frequency scale for the symptoms of GERD) at 2 week after double dose rabeprazole treatment

SECONDARY OUTCOMES:
sustained symptom improvement at 6 week after treatment | 6 weeks
  sustained symptom improvement assessed by FSSG(the frequency scale for the symptoms of GERD)score at 6 week after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tae Oh Kim, M.D. PhD., Study Director — Internal Medicine, Haeundae Paik Hospital; Eun Hee Seo, M.D, Principal Investigator — Internal Medicine, Haeundae Paik Hospital
Locations (1):
- Haeundae Paik Hospital, Inje University School of Medicine, Busan, South Korea